CLINICAL TRIAL: NCT04115761
Title: A Phase II, Randomized, Open-Label, Parallel-Group Study to Evaluate the Efficacy and Safety of Autologous Dendritic Cell Vaccination (ADCV01) As an Add-On Treatment for Primary Glioblastoma Multiforme (GBM) Patients
Brief Title: Evaluate the Efficacy and Safety of ADCV01 As an Add-On Treatment for Primary Glioblastoma Multiforme (GBM) Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ever Supreme Bio Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ES-CDCV01-A2201
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: GBM

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigational Group (Other): ADCV01 is autologous dendritic cells (DCs) stimulated by the patients' own tumor antigens. The total 10 doses (1 mL/dose; 2±0.5 × 10^7 cell/dose) of ADCV01 will be administered to patients assigned to the investigational group. The ADCV01 will be administered to the bilateral subaxillary subcutaneous regional lymph nodes (half of volume about 0.5 mL of ADCV01) once weekly for the first 4 doses, and the following 2 treatments will be administered bi-weekly. The last 4 treatments will be administered every 4 weeks.
  Interventions: Biological: autologous dendritic cells
- Control Group (Other): the conventional treatment (RT and chemotherapy) will be given after tumor resection, followed by subsequent evaluations by an approximately 8-week interval.
  Interventions: Biological: autologous dendritic cells

INTERVENTIONS:
Biological: autologous dendritic cells — The total 10 doses (1 mL/dose; 2±0.5 × 10^7 cell/dose) of ADCV01 will be administered to patients assigned to the investigational group. The ADCV01 will be administered to the bilateral subaxillary subcutaneous regional lymph nodes (half of volume about 0.5 mL of ADCV01) once weekly for the first 4 doses, and the following 2 treatments will be administered bi-weekly. The last 4 treatments will be administered every 4 weeks.

SUMMARY:
This study is designed with open-label and randomized parallel group to evaluate the efficacy and safety of autologous dendritic cell vaccination (ADCV01) as an add-on treatment for primary glioblastoma multiforme

DETAILED DESCRIPTION:
The patients with primary glioblastoma multiforme (GBM) have high mortality and morbidity. Even with best conventional therapy (surgery, radiation, and chemotherapy), the most of median survivals are less than 2 years. The one-year progression-free survival (PFS) is less than 20%. Recently, the immune therapy is a new promising therapy for GBM from the evidences of published experimental data and clinical trials.

However, the outcomes of immune therapy are still equivocal. The critical point of immune therapy is strongly influenced by tumor microenvironment. Up to now, for example, immune checkpoint inhibitor such as programmed cell death protein ligand 1 (PD-L1) and programmed cell death protein 1 (PD-1) was found to induce exhaustion of CD8 T cell by of PD-1/PD-L1 reaction. Unfortunately, GBM cells always have high PD-L1 expression. It means the higher PD-1 level of T-cell indicates the higher immune suppression by GBM tumor cells.

In the investigators preclinical study, the best murine survival was found to be the combination outcome of dendritic cell (DC) with anti-PD-1 therapy which was better than that of DC therapy only. From previously ADCV-treated patients, the median of PD-1/CD8 was 0.21. When the PD-1/CD8 ratio less than 0.21, this patient is defined as with low PD-1 level.

From the investigators previous experience, patients with low PD-1/CD8 ratio had far better 2-year overall survival (OS) than patients with high PD-1/CD8 ratio in ADCV treatment. On the other hand, it showed that OS and PFS had significant reverse correlation with PD-1 level of Tcell during DC immunotherapy. Considering the needs and benefit of patients, the new autologous dendritic cell vaccine (ADCV01) is proposed to be added on conventional therapy in low PD-1 expressed GBM patients and evaluate its safety and efficacy.

In this study, only newly diagnosed primary GBM (wild-type Isocitrate Dehydrogenase 1, IDH-1) patients will be enrolled in this clinical trial. In addition to fulfilling all inclusion criteria without matching any of the exclusion criteria, patients will undergo tumor resection and less than 25% of residual tumor size, followed by being subjected to histological analysis. Examinations of molecular diagnostics including IDH-1 for confirmation of IDH-1 wild-type GBM according to the 2016 WHO Classification of Tumors of the Central Nervous System, and cut-off criteria for expression levels of PD-1 and CD8 (PD-1/CD8 ratio less than 0.21) will be screened for the eligibility to participate in this study and MGMT status will also be determined.

After tumor resection, all eligible patients will receive standard radiotherapy (RT) plus Temozolomide (Temodal, TMZ), followed by adjuvant treatment of TMZ. Patients assigned to the investigational group will receive ADCV01 administration as an add-on treatment after operation in this study.

This study aims to treat eligible patients with ADCV01 as an add-on immunotherapy along with post-surgery GBM treatment and compare the treatment to the conventional therapy (RT plus standard TMZ chemotherapy) alone on the basis of PFS in an unbalanced allocation (investigational group : control group = 2:1). After tumor resection, patients assigned to the control group will receive RT plus TMZ, followed by the scheduled evaluation visits. For patients assigned to the investigational drug group, a standard of 10 doses of ADCV01 (2±0.5 × 10^7 cell/dose) in addition to conventional therapy will be administered.

The assessment of tumor response is based on [Update Response Assessment Criteria for High-Grade Gliomas, Response Assessment in Neuro-Oncology (RANO)] assessed by the on-site investigator and Blinded Independent Central Review (BICR) independently. If needed, the repeat operation for decompressive craniotomy evaluated by the on-site neurosurgeon for relief of increased intracerebral pressure (IICP), or for lifesaving will be allowed in both groups. However, in this study, the reoperation for recurrent tumor will be allowed.

RT will be given if feasible considering the total RT accumulatively given is not enough when tumor recurs (total dose 60 Gy). Gamma knife will not be used for recurrent tumor in this study which is different application from previous research.

Regardless of receiving re-operation or not in both groups, TMZ treatment will be shifted to anti-angiogenic therapy (AVASTIN®) 10 mg/kg/2weeks for 6 doses after patients have recurrence of GBM. Pseudo-progression may lead to either premature termination of therapy or unnecessary debulking surgeries. Therefore, adjuvant TMZ is recommended to be continued for a minimum of 3 cycles (along with ADCV01 treatment in the first 3 months of the adjuvant TMZ period), after which other imaging techniques (e.g., Gdenhancing MRI and proton magnetic resonance spectroscopy) should be used to ascertain progression. TMZ is not continuously used whenever recurrence. On this end, the treatment course is complete.

If the recurrent GBM in patients assigned to the investigational group is occurred before completing 10 doses of ADCV01 treatments, the patient will be treated by the remaining ADCV01 and complete the originally scheduled treatment.

In this phase II study, 24 eligible primary GBM patients who are with low PD-1/CD8 ratio will be recruited. There will be 16 patients with combination of ADCV01 and conventional therapy, and 8 patients with conventional therapy only. In this trial, the treatment efficacy of ADCV01 measured by one-year PFS rate will be evaluated at the end of phase II study. Because PFS was surrogate endpoint of overall survival in GBM by literature-based meta-analysis from 91 clinical trials, the 1-year PFS rate will be the primary endpoint of GBM clinical trial.

This study is designed with open-label and randomized parallel group. To date, 34 clinical trials of DC for GBM published up to 2017 in ClinicalTrials.gov, there are 5/34 trials designed by double blinded method and 2/34 trials by single blinded and most of 27/34 trials by open-label (please see ref. ClinicalTrials.gov). The other reason for open-label is that the apheresis for control patients is an invasive procedure. GBM is a not easily curable disease; patients with MGMT methylation have a better survival than with unmethylation. In this trial, MGMT status will be evaluated in all tumor specimens for further subgroup analysis.

ELIGIBILITY:
Inclusion Criteria:

Stage I (Pre-screening)

1. Patients are ≥ 20 and ≤ 75 years of age at brain tumor resection surgery.
2. Patients with newly diagnosed single, primary, WHO grade IV, glioblastoma (except for locating on brainstem or cerebellum) scheduled to undergo craniotomy tumor excision, and are willing to preserve the resected tumor cells enabling the production of ADCV01.
3. Patients undergo tumor resection by aid of neuro-navigation without receiving any intracranial implantation therapies (e.g., BCNU wafer).
4. Only one GBM tumor number.
5. Patients must be able to understand and sign the informed consent documents and aware of the investigational nature of the study.
6. Patients have the expected life expectancy of > 12 weeks at the pre-screening visit as judged by the investigator.
7. Patients with stable vital sign and KPS ≥ 70 at the pre-screening visit.
8. Patients with adequate renal function at the pre-screening visit:

   serum creatinine < 1.8 mg/dL; creatinine clearance > 30 mL/min
9. Patients with adequate liver function at the pre-screening visit:

   AST, ALT, and ALP ≤ 3× upper limit of normal (ULN); and total bilirubin < 3 mg/dL
10. Patients with prothrombin time and activated partial thromboplastin time ≤ 1.5× ULN at the pre-screening visit
11. Patients with adequate hematopoietic function at the prescreening and before administration of study medication

    1. Absolute neutrophil count (ANC) ≥ 1,000 cells/μL
    2. Platelets ≥ 100,000 counts/μL
    3. Total white blood cell (WBC) ≥ 2,000 cells/μL
    4. Hemoglobin ≥ 8 g/dL
12. All male and female patients with child-bearing potential (between puberty and 2 years after menopause) must be practicing sexual abstinence and be willing to continue to use a medically acceptable form of birth control for at least 1 month prior to screening (that period will extend to 3 months for oral contraceptive use). The patients should use appropriate contraceptive method(s) as shown below, until at least 6 months after the last dose of ADCV01 administration.

    1. Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, thermal symptom post-ovulation methods) and withdrawal are not acceptable methods of ontraception).
    2. Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least 6 weeks before administration of study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
    3. Male sterilization (at least 6 months prior to screening). For female subjects in the study, the vasectomized male partner should be the sole partner for that subject
    4. Combination of any two of the following listed methods:

    (d.1+d.2 or d.1+d.3, or d.2+d.3): d.1 Use of oral, injected, or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception. d.2 Placement of an intrauterine device (IUD) or intrauterine system (IUS). d.3 Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository.
13. Patients agree to be in compliance with treatment plan as planned in the clinical protocol.

    Stage II (Screening/Randomization) In addition to fulfill the criteria in Stage I, following criteria should be met to be eligible for remaining in the study.
14. Patients' resected brain tumors are pathologically confirmed cases of the IDH-1 wild-type glioblastoma, and patients are willing to do monocyte-collecting apheresis at the screening/randomization visit.
15. At the screening/randomization visit, patients' resected brain tumors are confirmed of low PD-1+/ CD8+ ratio (ratio <0.21).
16. Residual tumor with less than 25% contrast-enhancing mass on post-surgical brain MRI (within 2 days post-operation) as assessed by the neurosurgeon and/or radiologist.

Exclusion Criteria:

Stage I (Pre-screening)

1. Number of GBM is more than one
2. Patient who has participated in other investigational studies within 4 weeks prior to pre-screening
3. Patient with known or suspected hypersensitivity to ADCV01 or its excipients
4. Patient who has a history of hypersensitivity reaction (e.g., urticarial, allergic reaction including anaphylaxis, toxic epidermal necrosis, and Stevens-Johnson syndrome) to dacarbazine (DTIC) or any components of medications of temozolomide and bevacizumab
5. Patient has acute infectious disease or acute cardiovascular disease; clinically manifest myocardial insufficiency or history of myocardial infarction during the past 6 months prior to prescreening; or has active uncontrolled arterial hypertension as supported by medical history.
6. Patient has clinically significant immuno-compromised condition (other than that related to the use of corticosteroids), is human immunodeficiency virus positive (anti-HIV and nucleic acid test) or medical condition requiring systemic immunesuppressive treatments.
7. Patient with active rheumatic disease or other collagen vascular disease, or is with active autoimmune disorder or known history of an autoimmune neurologic condition (e.g., Guillain-Barre syndrome). Patients with vitiligo, type 1 diabetes mellitus, hypothyroidism due to autoimmune condition, only requiring hormone replacement therapy are permitted to enroll.
8. Patients with psoriasis requiring systemic therapy, or conditions expected to recur in the presence of an external trigger
9. Patient with syphilis, acute HBV, HCV (except hepatitis carriers), HTLV-I/II, CMV, or an increased risk (or has been diagnosed) for human transmissible spongiform encephalopathy (TSE); including Creutzfeldt-Jakob disease (CJD)
10. Patient with history of coagulation disorder associated with bleeding or recurrent thrombotic events
11. Patient with medical, social, or psychological factors interfering with compliance of the study
12. Female patient who is lactating, pregnant, or planned to be pregnant
13. Inability to undergo MRI for any reason
14. History of malignancy other than glioma that is not stable in the past 5 years prior to pre-screening (informed consent form signing date)
15. Patient not suitable to participate the trial as judged by the investigator. Stage II (Screening/Randomization)

    The patient will be no longer eligible to participate the study if he/she met any of the following criteria:
16. GBM patients with high PD-1+/CD8+ ratio ≥ 0.21
17. GBM patients with mutant IDH-1
18. Residual tumor volume more than 25% of pre-operative tumor size.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-06-06 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
One-year progression-free survival (PFS) rate | the percentage of patients surviving 1 year after randomization without objective tumor progression or death.
  The PFS is defined as the time from randomization until the tumor objective progression or death, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Liang Huang, Study Director — Ever-Supreme Biotechnology
Locations (3):
- Taiwan (3):
  - Taichung Veterans General Hospital, Taichung, Non-US
  - Chang-Gung Memorial Hospital at Lin-Ko, Taoyuan District, Non-US
  - China Medical University Hospital, Taichung

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jan CI, Tsai WC, Harn HJ, Shyu WC, Liu MC, Lu HM, Chiu SC, Cho DY. Predictors of Response to Autologous Dendritic Cell Therapy in Glioblastoma Multiforme. Front Immunol. 2018 May 29;9:727. doi: 10.3389/fimmu.2018.00727. eCollection 2018. PMID 29910795
- [Background] Han K, Ren M, Wick W, Abrey L, Das A, Jin J, Reardon DA. Progression-free survival as a surrogate endpoint for overall survival in glioblastoma: a literature-based meta-analysis from 91 trials. Neuro Oncol. 2014 May;16(5):696-706. doi: 10.1093/neuonc/not236. Epub 2013 Dec 12. PMID 24335699
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009